CLINICAL TRIAL: NCT00314119
Title: Natural History and Biology of Dermal Neurofibromas in Neurofibromatosis Type 1
Brief Title: Natural History and Biology of Skin Neurofibromas in Neurofibromatosis Type 1
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060134; 06-C-0134
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-07-14

CONDITIONS: Neurofibromatosis Type 1; Neurofibroma
Keywords: Tumor Imaging; NF1; Natural History; Neurofibromatosis
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma; Neurofibromatoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Men and women between 20 and 50 years of age diagnosed with NF1 and their biological parents are eligible for this study.

SUMMARY:
This study will explore the growth of dermal neurofibromas (skin tumors) in patients with neurofibromatosis type 1 (NF1). Investigators will try to learn: 1) how fast (or slow) these benign tumors grow in NF1, 2) how often new tumors appear and 3) what genes are involved in the growth of the tumors.

Men and women between 20 and 50 years of age diagnosed with NF1 and their biological parents are eligible for this study.

Patients with NF1 are evaluated at the NIH Clinical Center with the following tests and procedures:

* Medical examination and drawing of family tree.
* Photos of the back, abdomen and thigh in order to count the number of skin tumors.
* Photos of the skin taken with a special camera (Primos camera) that takes very detailed pictures of a small area of skin.
* Photos of the skin taken with a dermatoscope, which takes very detailed pictures of a small area of skin under high magnification.
* Biopsy of at least one skin tumor and biopsy of a small piece of normal skin.
* Blood sample collection for genetic testing of the gene NF1 and to establish a cell line.
* Other medical tests (e.g., x-rays or MRI) if needed.

Patients and their families will also have a genetic counseling session and an opportunity to ask questions about neurofibromatosis type 1.

Patients return to the NIH after 3, 6, 12, 18 and 24 months for follow-up photographs and possibly blood samples.

Biological parents of patients provide a blood sample for genetic testing.

DETAILED DESCRIPTION:
This protocol results from a funded 2005 Bench-to-Bedside Award and explores the genetic basis of disease severity in neurofibromatosis type 1 (NF1) and the evaluation of three methods to measure disease progression of dermal neurofibromas. NF1 is a common multisystem genetic disorder associated with the development of benign and malignant tumors, primarily of the nervous system. NF1 is 100% penetrant and features variable expressivity and limited phenotype/genotype correlation. No standard treatment other than surgery exists for most NF1-associated tumors. Many aspects of the natural history of NF1-associated tumors are not fully characterized and require investigation to assess the effects of potential new treatments, in future clinical trials. The development of medical treatments for NF1-associated tumors is an important goal given their morbidity and the lack of non-surgical treatment options. The ability to predict the ultimate severity of disease would have a significant impact on the management and treatment of individuals with NF1.

Sorafenib (BAY 43-9006) is a novel, orally bioavailable agent that targets downstream effectors in the Ras signaling pathway (a key dysregulated pathway in NF1). It has thus a strong scientific rationale for evaluation in NF1 related tumors. Dermal neurofibromas occur in nearly every individual with NF1, and are a significant cosmetic problem and a major cause of morbidity. This protocol will 1) quantify the growth of dermal neurofibromas in NF1 with 3 different imaging modalities 2) use an innovative gene expression method to identify genetic modifiers of dermal neurofibroma burden, and 3) evaluate dermal neurofibromas and normal skin for the presence of targets of sorafenib. Successful validation of reliable quantitative imaging methods of dermal neurofibroma growth is a logical prerequisite to subsequent clinical trials with medical treatments, which will evaluate the effect of new agents on the growth rate of dermal neurofibromas. Identification of genetic modifiers may permit prediction of ultimate tumor burden. Evaluation of targets of new agents in dermal neurofibromas will allow for more rationale drug development for NF1. Given the paucity of protocols for adults with NF1 and dermal neurofibromas, this study will likely generate great interest among affected individuals and have rapid accrual.

ELIGIBILITY:
-INCLUSION CRITERIA - GROUP A INDIVIDUALS:

1. Clinical diagnosis of NF1. In order to meet the diagnosis of NF1 individuals must have 2 of the diagnostic criteria listed below:

   * Six or more cafe-au-lait macules (greater than or equal to 0.5 cm in prepubertal subjects or greater than or equal to 1.5 cm in postpubertal subjects)
   * Freckling in the axilla or groin
   * A tumor of the optic pathway
   * Two or more Lisch nodules
   * A distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
   * A plexiform neurofibroma or two or more neurofibromas
   * A first-degree relative with NF1 by the above criteria

   We may request the medical records of potential enrollees for our review. Ideally, individuals will have been evaluated by a geneticist and a definitive diagnosis made. However given the unique, familial (and often unmistakable features) of NF1 it is likely the diagnosis can be reliably made by a non-geneticist.
2. Age at study entry: 20- 50 years (inclusive)
3. Identification of a physician who will be responsible for follow-up care, if needed
4. Ability and willingness to travel to the NIH Clinical Center or University of Alabama at Birmingham Alabama for multiple evaluations
5. Ability and willingness of both biologic parents to provide a blood (or saliva) sample
6. Must have at least one dermal neurofibroma amenable to excisional biopsy. Preferably the neurofibroma will be on the thorax or abdomen and be at least the size of a pencil eraser.

INCLUSION CRITERIA - GROUP B INDIVIDUALS:

1. Biological parents (either affected or unaffected) of Group A individuals
2. Willingness to donate a blood or saliva sample for genotyping
3. Willing to undergo a brief skin and eye exam at the NIH CC (to rule out NF1) or University of Alabama, if accompanying adult children

EXCLUSION CRITERIA - GROUP A INDIVIDUALS

MEDICAL INCLUSIONS:

1. Any history of administration (or current use) of radiation therapy, chemotherapeutic agents or biologic agents (experimental or not) that resulted in a documented significant change in dermal neurofibroma tumor burden or growth.
2. Patients with probable segmental or mosaic NF1 will be excluded from study participation and medical records may be reviewed prior to enrollment for this determination.
3. A history of administration of medications within 6 months of study entry that might reasonably be expected to alter the natural history of tumor growth (examples include pirfenidone, interferon, farnesyl transferase inhibitor (FTI), MTX/VBL, thalidomide, growth hormone) or cause significant changes in gene expression profile.
4. Known or suspected untreated bleeding diathesis or platelet disorder that would preclude safe and successful dermal neurofibroma and skin biopsy. Patients prescribed aspirin or other known/suspected agent that interferes with platelet function may also be excluded if they cannot safely discontinue its use a week ahead of the biopsy.
5. Clinically significant unrelated systemic illness, such as serious infection, hepatic, renal or other organ dysfunction, which in the judgment of the principal investigator or associate investigator would compromise the patient's ability to participate in the study procedures.
6. Inability or unwillingness to tolerate the dermal neurofibroma excision and skin biopsy or blood draw.

VULNERABLE POPULATIONS EXCLUSIONS

1) Cognitive delay to the extent that conscious sedation is required to obtain the dermal neurofibroma excision and skin biopsy.

OTHER EXCLUSIONS

1. Biologic parents unable or unwilling to provide a blood (or saliva) sample.
2. Inability to travel to the NIH or to The University of Alabama at Birmingham, AL
3. Individuals refusing an excisional tumor or skin biopsy.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women between 20 and 50 years of age diagnosed with NF1 and their biological parents are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2006-06-08 (Actual)

PRIMARY OUTCOMES:
Quantify the growth of dermal neurofibromas in NF1 with 3 different imaging modalities. | 12/31/2010
  Evaluate the natural history of dermal neurofibromas in NF1 by monitoring the growth rate and development of new dermal neurofibromas using three different complementary imaging modalities over time in individuals with NF1. The study will be adequately powered so that a minimally meaningful statistical definition of progression can be developed for use in subsequent treatment protocols.
Use an innovative gene expression method to identify genetic modifiers of dermal neurofibroma burden. | 12/31/2010
  Screen for genetic modifiers of dermal neurofibroma burden and growth using a novel approach employing the genetics of gene expression and family-based tests of association. Characterization of gene expression profiles in lymphoblastoid cell lines (LCLs) and dermal neurofibromas predictive of tumor behavior (e.g. growth rate) will also be explored.
Evaluate dermal neurofibromas and normal skin for the presence of targets of sorafenib. | 12/31/2010
  Validate sorafenib as a rational agent for clinical development in individuals with NF1-related dermal neurofibromas. Quantify thelevel of expression of the targets of sorafenib by gene expression microarray of both normal skin and of the dermal neurofibromasthemselves. A tissue microarray from formalin-fixed neurofibromas may also be developed to investigate the expression of other therapeutic targets.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Stewart, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical data will be shared with collaborators under appropriate agreements.
Supporting Information: Study Protocol
Time Frame: At the time of a request and as long as needed.
Access Criteria: De-identified clinical data will be shared with collaborators under appropriate agreements.

REFERENCES:
- [Background] Korf BR. Clinical features and pathobiology of neurofibromatosis 1. J Child Neurol. 2002 Aug;17(8):573-7; discussion 602-4, 646-51. doi: 10.1177/088307380201700806. PMID 12403555
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-C-0134.html